CLINICAL TRIAL: NCT03181386
Title: Prospective Study of the Assessment of the Dental Protocol for Tooth Extraction in Patients With Atrial Fibrillation in Continuous Use of New Oral Anticoagulants: A Pilot Study
Brief Title: Tooth Extraction in Patients With Atrial Fibrillation in Use of New Oral Anticoagulants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Itamara Lucia Itagiba Neves, PhD, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Odonto-NOAC
Record Dates: First submitted 2017-06-02; First posted 2017-06-08 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation; Periodontal Disease; Hemorrhage
Keywords: Dabigatran; Rivaroxaban; Apixaban; Warfarin; Tooth Extraction
MeSH Terms: conditions — Atrial Fibrillation; Periodontal Diseases; Hemorrhage | interventions — Rivaroxaban; Dabigatran; apixaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rivaroxaban (Experimental): As the rivaroxaban is ingested 1x/day, the interval between a maximum peak concentration and the other peak is 24 hours. Therefore, the surgery will be performed between two peaks of maximum drug concentration, knowing that the maximum peak concentration is an average of two hours after ingestion. So the surgical procedure should be scheduled 14 hours (2 hours+ 12 hours) after the last medication intake.
  Interventions: Drug: Rivaroxaban
- Dabigatran and Apixaban (Experimental): As dabigatran and apixaban are taken 2x/day, the interval between two peak concentration is 12 hours.Taking into account the first two hours of maximum peak concentration and half the interval between two peaks (2 hours + 6 hours = 8 hours), the surgical procedure must be programmed eight hours after the last intake of medication.
  Interventions: Drug: Dabigatran and Apixaban
- Warfarin (Active Comparator): The control group will consist of patients on chronic use of warfarin. The operation will be scheduled at any time, provided that the patient has INR value between 2.0 and 3.0 and test performed in maximum 15 days before surgery.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 15 or 20mg tablet by mouth, every 24 hours, continuous use.
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Dabigatran and Apixaban — Dabigatrana 110 or 150 mg tablet and Apixaban 2,5 or 5mg tablet by mouth, every 12 hours, continuous use.
  Other Names: Pradaxa and Eliquis
  Arms: Dabigatran and Apixaban
Drug: Warfarin — The dosage of Warfarin is individualized for each patient, according to the patient's TP/INR value. The value of TP/INR should be in the therapeutic dosage of 2.0 to 3.0
  Other Names: Marevan
  Arms: Warfarin

SUMMARY:
The purpose of this study is to evaluate the safety of a protocol which does not suspend the new oral anticoagulants (dabigatran, rivaroxaban and apixaban) in front of dental extractions in patients with non-valvular atrial fibrillation.

DETAILED DESCRIPTION:
The sample will be divided into three groups according to the pharmacokinetics of the oral anticoagulant: rivaroxaban 1x/day (group 1); dabigatran and apixabana 2x/day (group 2) and warfarin (control group). Extraction of one to three teeth will be scheduled, in the valley of the new oral anticoagulants' concentration, considered the period of smallest haemorrhagic risk without suspension. In group 1 the surgery will be scheduled 14 hours after the last intake, in group 2 the surgery will be scheduled 8 hours after the last intake, while the control group will undergo the procedure with INR values between 2.0 and 3,0. Hemostatic measures with tranexamic acid paste intra alveolar, suture and biological glue GRF® (gelatin, resorcinol and formaldehyde) and post operative care will be associated. The patients will be contacted after the procedure to inform the presence or absence of late bleeding. The patient should return 24 hours later to evaluate the surgical site. This protocol is based on Guidelines and scientific articles, pharmacokinetics and clinical experience of the authors.

ELIGIBILITY:
Inclusion Criteria:

* Selection of patients: Both genders, aged over 18 years, regardless of ethnicity, marital status, nationality, naturalness or profession, with non-valvular atrial fibrillation using dabigatran or rivaroxaban or apixaban or warfarin, under medical outpatient treatment or during the hospitalization period.
* Dentistry: Patients with indications of exodontia of one to three permanent adjacent teeth erupted in the maxilla or mandible due to extensive dental caries or periodontal disease.

Exclusion Criteria:

* Clinical: Patients on concomitant use of antiplatelet agents or heparin, pregnant and lactating patients, with coagulation disorders, severe chronic renal insufficiency (CrCl <30), severe hepatopathies and proven to be allergic to lidocaine and / or epinephrine.
* Dentistry: Odontophobic, edentulous, or healthy teeth; Deciduous teeth and Included teeth.
* Regarding the time of medication intake: Regarding the time of medication intake Patients taking rivaroxaban who routinely take the medication between 5:00 a.m. to 4:00 p.m. (unworkable schedule for surgery) that do not accept a change in the intake schedule suggested by the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
A bleeding event (incidence of postoperative bleeding events) | 7 days
  To evaluate the safety of a protocol regarding the risks of bleeding after dental extractions performed in patients with non-valvular atrial fibrillation in continuous use of the new oral anticoagulants, we compared the incidence of postoperative bleeding events after dental extractions between patients in use of new oral anticoagulants and those treated of warfarin without withdrawal of oral anticoagulant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Denise T Hachul, PhD, Study Director — Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo; Itamara LI Neves, PhD, Principal Investigator — Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo; Elaine M Higashi, S, Study Chair — Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo; Ricardo S Neves, PhD, Study Chair — Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo; Francisco CC Darrieux, PhD, Study Chair — Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo; Mauricio I Scanavacca, PhD, Study Chair — Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After thesis defense, the IPD will be available on the Portal Digital Library of Theses and Dissertations of the University of São Paulo (http://www.teses.usp.br/index.php?option=com_jumi&fileid=12&Itemid=77&lang=ptbr), in a PDF file.

REFERENCES:
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Background] Fakhri HR, Janket SJ, Jackson EA, Baird AE, Dinnocenzo R, Meurman JH. Tutorial in oral antithrombotic therapy: biology and dental implications. Med Oral Patol Oral Cir Bucal. 2013 May 1;18(3):e461-72. doi: 10.4317/medoral.19140. PMID 23524440
- [Background] Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH; ESC Committee for Practice Guidelines. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Europace. 2010 Oct;12(10):1360-420. doi: 10.1093/europace/euq350. No abstract available. PMID 20876603
- [Background] Halvorsen S, Atar D, Yang H, De Caterina R, Erol C, Garcia D, Granger CB, Hanna M, Held C, Husted S, Hylek EM, Jansky P, Lopes RD, Ruzyllo W, Thomas L, Wallentin L. Efficacy and safety of apixaban compared with warfarin according to age for stroke prevention in atrial fibrillation: observations from the ARISTOTLE trial. Eur Heart J. 2014 Jul 21;35(28):1864-72. doi: 10.1093/eurheartj/ehu046. Epub 2014 Feb 20. PMID 24561548
- [Background] Little JW. New oral anticoagulants: will they replace warfarin? Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 May;113(5):575-80. doi: 10.1016/j.oooo.2011.10.006. Epub 2012 Mar 3. PMID 22668618
- [Background] Firriolo FJ, Hupp WS. Beyond warfarin: the new generation of oral anticoagulants and their implications for the management of dental patients. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Apr;113(4):431-41. doi: 10.1016/j.oooo.2011.10.005. PMID 22668425
- [Background] Elad S, Marshall J, Meyerowitz C, Connolly G. Novel anticoagulants: general overview and practical considerations for dental practitioners. Oral Dis. 2016 Jan;22(1):23-32. doi: 10.1111/odi.12371. Epub 2015 Nov 16. PMID 26386350
- [Background] van Ryn J, Stangier J, Haertter S, Liesenfeld KH, Wienen W, Feuring M, Clemens A. Dabigatran etexilate--a novel, reversible, oral direct thrombin inhibitor: interpretation of coagulation assays and reversal of anticoagulant activity. Thromb Haemost. 2010 Jun;103(6):1116-27. doi: 10.1160/TH09-11-0758. Epub 2010 Mar 29. PMID 20352166
- [Background] Romond KK, Miller CS, Henry RG. Dental management considerations for a patient taking dabigatran etexilate: a case report. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Sep;116(3):e191-5. doi: 10.1016/j.oooo.2013.05.001. Epub 2013 Jul 10. PMID 23850368
- [Background] Davis C, Robertson C, Shivakumar S, Lee M. Implications of Dabigatran, a direct thrombin inhibitor, for oral surgery practice. J Can Dent Assoc. 2013;79:d74. PMID 23920075
- [Background] Turpie AG, Kreutz R, Llau J, Norrving B, Haas S. Management consensus guidance for the use of rivaroxaban--an oral, direct factor Xa inhibitor. Thromb Haemost. 2012 Nov;108(5):876-86. doi: 10.1160/TH12-03-0209. Epub 2012 Sep 26. PMID 23014816
- [Background] Weinz C, Schwarz T, Kubitza D, Mueck W, Lang D. Metabolism and excretion of rivaroxaban, an oral, direct factor Xa inhibitor, in rats, dogs, and humans. Drug Metab Dispos. 2009 May;37(5):1056-64. doi: 10.1124/dmd.108.025569. Epub 2009 Feb 5. PMID 19196845
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Haas S, Bode C, Norrving B, Turpie AG. Practical guidance for using rivaroxaban in patients with atrial fibrillation: balancing benefit and risk. Vasc Health Risk Manag. 2014 Mar 10;10:101-14. doi: 10.2147/VHRM.S55246. eCollection 2014. PMID 24648742
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Friedman RJ, Kurth A, Clemens A, Noack H, Eriksson BI, Caprini JA. Dabigatran etexilate and concomitant use of non-steroidal anti-inflammatory drugs or acetylsalicylic acid in patients undergoing total hip and total knee arthroplasty: no increased risk of bleeding. Thromb Haemost. 2012 Jul;108(1):183-90. doi: 10.1160/TH11-08-0589. Epub 2012 May 3. PMID 22552763
- [Background] Hartter S, Sennewald R, Schepers C, Baumann S, Fritsch H, Friedman J. Pharmacokinetic and pharmacodynamic effects of comedication of clopidogrel and dabigatran etexilate in healthy male volunteers. Eur J Clin Pharmacol. 2013 Mar;69(3):327-39. doi: 10.1007/s00228-012-1304-8. Epub 2012 Jul 11. PMID 22782539
- [Background] Kubitza D, Becka M, Mueck W, Zuehlsdorf M. Safety, tolerability, pharmacodynamics, and pharmacokinetics of rivaroxaban--an oral, direct factor Xa inhibitor--are not affected by aspirin. J Clin Pharmacol. 2006 Sep;46(9):981-90. doi: 10.1177/0091270006292127. PMID 16920892
- [Background] Eriksson BI, Rosencher N, Friedman RJ, Homering M, Dahl OE. Concomitant use of medication with antiplatelet effects in patients receiving either rivaroxaban or enoxaparin after total hip or knee arthroplasty. Thromb Res. 2012 Aug;130(2):147-51. doi: 10.1016/j.thromres.2011.12.005. Epub 2012 Jan 5. PMID 22225858
- [Background] Scott A, Gibson J, Crighton A. The management of dental patients taking new generation oral anticoagulants. Prim Dent J. 2014 Nov;3(4):54-8. doi: 10.1308/205016814813877289. PMID 25668377
- [Background] Heidbuchel H, Verhamme P, Alings M, Antz M, Hacke W, Oldgren J, Sinnaeve P, Camm AJ, Kirchhof P; European Heart Rhythm Association. European Heart Rhythm Association Practical Guide on the use of new oral anticoagulants in patients with non-valvular atrial fibrillation. Europace. 2013 May;15(5):625-51. doi: 10.1093/europace/eut083. PMID 23625942
- [Background] Hong C, Napenas JJ, Brennan M, Furney S, Lockhart P. Risk of postoperative bleeding after dental procedures in patients on warfarin: a retrospective study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Oct;114(4):464-8. doi: 10.1016/j.oooo.2012.04.017. PMID 22986241
- [Background] Sie P, Samama CM, Godier A, Rosencher N, Steib A, Llau JV, Van der Linden P, Pernod G, Lecompte T, Gouin-Thibault I, Albaladejo P; Working Group on Perioperative Haemostasis; French Study Group on Thrombosis and Haemostasis. Surgery and invasive procedures in patients on long-term treatment with direct oral anticoagulants: thrombin or factor-Xa inhibitors. Recommendations of the Working Group on Perioperative Haemostasis and the French Study Group on Thrombosis and Haemostasis. Arch Cardiovasc Dis. 2011 Dec;104(12):669-76. doi: 10.1016/j.acvd.2011.09.001. Epub 2011 Oct 29. PMID 22152517
- [Background] Clemm R, Neukam FW, Rusche B, Bauersachs A, Musazada S, Schmitt CM. Management of anticoagulated patients in implant therapy: a clinical comparative study. Clin Oral Implants Res. 2016 Oct;27(10):1274-1282. doi: 10.1111/clr.12732. Epub 2015 Nov 23. PMID 26592859